CLINICAL TRIAL: NCT06438497
Title: The Effect of Different Body Positions and Channel Sheaths on Retrograde Intrarenal Stone Surgery(RIRS) Treatment of Lower Pole Renal Stones: a Randomized Controlled Trial
Brief Title: The Effect of Different Body Positions and Channel Sheaths on RIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(84)2024
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Urolithiasis
Keywords: RIRS; lower pole renal stones; stone-free rate; ureteral access sheath; flexible negative-pressure; lateral position
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RIRS with f-UAS, lateral position (Experimental): In group 1, patients were placed on operating table in lateral position. A flexible negative-pressure suction ureteric access sheath (f-UAS) is placed under the pelvi-ureteral junction (PUJ) in RIRS.
  Interventions: Procedure: RIRS with f-UAS, lateral position
- RIRS with f-UAS, lithotomy position (Experimental): In group 2, patients were placed on operating table in lithotomy position. A flexible negative-pressure suction ureteral access sheath (f-UAS) is placed under the pelvi-ureteric junction (PUJ) in RIRS.
  Interventions: Procedure: RIRS with f-UAS, lithotomy position
- RIRS with traditional UAS, lateral position (Experimental): In group 3, patients were placed on operating table in lateral position. A traditional ureteric access sheath (UAS) is placed under the pelvi-ureteral junction (PUJ) in RIRS.
  Interventions: Procedure: RIRS with traditional UAS, lateral position
- RIRS with traditional UAS, lithotomy position (Active Comparator): In group 4, patients were placed on operating table in lithotomy position. A traditional ureteral access sheath (UAS) is placed under the pelvi-ureteric junction (PUJ) in RIRS.
  Interventions: Procedure: RIRS with traditional UAS, lithotomy position

INTERVENTIONS:
Procedure: RIRS with f-UAS, lateral position — In this intervention, patients were placed on operating table in lateral position. The coronal plane of the patient body was perpendicular to the operating table. The upper limbs were extended and fxed with brackets. A f-UAS is placed under the pelvi-ureteric junction (PUJ) in RIRS. The tip of the UAS has good flexibility and deformability. It can passively bend with the bending of the flexible ureteroscope (f-URS).
  Arms: RIRS with f-UAS, lateral position
Procedure: RIRS with f-UAS, lithotomy position — In this intervention, patients were placed on operating table in lithotomy position. This position is common and standard. A f-UAS is placed under the pelvi-ureteric junction (PUJ) in RIRS. The tip of the UAS has good flexibility and deformability. It can passively bend with the bending of the flexible ureteroscope (f-URS).
  Arms: RIRS with f-UAS, lithotomy position
Procedure: RIRS with traditional UAS, lateral position — In this intervention, patients were placed on operating table in lateral position. The coronal plane of the patient body was perpendicular to the operating table. The upper limbs were extended and fxed with brackets. A traditional UAS is placed under the pelvi-ureteric junction (PUJ) in RIRS.
  Arms: RIRS with traditional UAS, lateral position
Procedure: RIRS with traditional UAS, lithotomy position — In this intervention, patients were placed on operating table in lithotomy position. This position is common and standard. A traditional UAS is placed under the pelvi-ureteric junction (PUJ) in RIRS.
  Arms: RIRS with traditional UAS, lithotomy position

SUMMARY:
Retrograde flexible ureteroscopy (RIRS) is currently the first-line treatment for renal stones < 2cm. Lower pole renal stones(LPS) are a difficult problem for urologists. The flexible negative pressure suction ureteral sheath(f-UAS) can facilitate RIRS to flush out the fragments and dust in time, and provide a clear vision and reduce the renal pelvis pressure(RPP) during operation.Standard lithotomy position is the most commonly used position for RIRS. Besides, T-tilt position is also available for RIRS in special cases. Investigators were inspired by this and proposed the lateral position, which is available in cases of LPS.In long-term practice, investigators have found that the change of position and the use of f-UAS can improve stone-free rate(SFR). Investigators aimed to conduct a prospective randomized controlled trial to compare the SFR of different positions and different ureteral sheaths.

DETAILED DESCRIPTION:
Urolithiasis was one of the most frequently noted diseases in urology clinic, with an incidence ranged from 5 to 15% around the world. Retrograde flexible ureteroscopy (RIRS) is currently the first-line treatment for renal stones < 2cm in size. Lower pole renal stones(LPS) are a difficult problem for urologists. The inborn sharp infundibular-pelvic angle (IPA) designated an inferior stone-free rate(SFR) of 65-82.5% in LPS when compared to middle and/or upper pole stone. The flexible negative pressure suction ureteral sheath(f-URS) can facilitate RIRS to flush out the fragments and dust in time, and provide a clear vision and reduce the renal pelvis pressure(RPP) during operation. Therefore, in cases of LPS, f-URS combined with RIRS may show advantages. However, there is currently a lack of relevant prospective randomized controlled studies. Standard lithotomy position is the most commonly used position for RIRS. Besides the standard lithotomy position, other positions, such as the T-tilt position, are also available for RIRS in special cases. Investigators were inspired by this and proposed the lateral position, which is available for RIRS in cases of LPS.Theoretically, in standard lithotomy position, the renal pelvis and renal calyces were mostly distributed in a '-<' shaped structure on the horizontal plane. However, the renal pelvis and renal calyxes would be stood up in a 'Y'-shaped structure when patients laid in lateral position. And gravity will make the calyceal stones at the dome fall into the renal pelvis naturally during the lithotripsy. In long-term clinical practice, researchers have found that the change of position and the use of f-UAS can improve SFR. The investigators aimed to conduct a prospective randomized controlled trial to compare the SFR of different positions and different ureteral sheaths.

ELIGIBILITY:
Inclusion Criteria:

* LPS with a diameter of 10-20 mm
* American Society of Anesthesiologists(ASA) score Ⅰ,Ⅱ and Ⅲ
* Adult patients

Exclusion Criteria:

* Ureteric stricture
* Urethral deformity
* Renal malformation, including horseshoe kidney, ectopic kidney and transplanted kidney
* Pregnancy
* Multiple stones in diferent calyces, including upper pole and middle pole

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | 1 day
  A low-dose and ultrathin 2-mm spiral CT was performed at 1 day postoperatively for evaluation of fnal SFR. Stone-free status was defined as no fragments observed or clinically insignifcant residual fragments (CIRF)<2 mm.
Stone-free rate | 1 month
  A low-dose and ultrathin 2-mm spiral CT was performed at 1 month postoperatively for evaluation of fnal SFR. Stone-free status was defined as no fragments observed or clinically insignifcant residual fragments (CIRF)<2 mm.

SECONDARY OUTCOMES:
Operative time | During surgery
  Surgery duration, minutes
Hemoglobin drop | 1 day after surgery
  Change of hemoglobin level 1 day after surgery comparing to pre-operative value, g/L
Hospital stay | 1 week
  Duration of hospital stay after surgery, days
Complication rate | 1 month after sugery
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.The investigator will invaluate perioperative complications by modified Clavien system

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China